CLINICAL TRIAL: NCT04429204
Title: Evaluation of Cryo-Immune Stimulation in Mesothelioma
Brief Title: Cryoablation for the Promotion of Local Tumor Infiltration in Patients With Mesothelioma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not opened
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-001175; NCI-2020-00640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-001175 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Basic science (cryoablation, tissue collection) (Experimental): At the time of standard of care pleural biopsy, patients undergo cryoablation over 30 minutes, then a sample of tissue from the ablated region and a non-ablated (tumor negative control) region are collected.
  Interventions: Procedure: Biospecimen Collection; Procedure: Cryosurgery

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tissue
Procedure: Cryosurgery — Undergo cryoablation
  Other Names: Ablation, Cryo; Cryoablation; cryosurgical ablation

SUMMARY:
This trial evaluates if cryoablation will stimulate a local immune response by cluster of differentiation 8 positive (CD8+) cells which are not present in ablation naive regions of the tumors in patients with mesothelioma. Cryoablation uses extreme cold to damage or destroy tumor lesions. Mesothelioma is a rare cancer that grows and spreads quickly, and has low survival rates. The information learned from this study may provide evidence as to whether there is a measurable, local immune response from cryoablation. Studying samples of mesothelioma tissue in the laboratory from patients who have undergone biopsy may help doctors learn more about the effects of cryoablation on cells. It may also help doctors understand how well patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the simple hypothesis that cryoablation of mesothelioma will promote local tumor infiltration by cytotoxic cluster of differentiation 8 positive (CD8+) cells that will not be present in ablation naive regions of the tumors.

II. To determine whether there is a preponderance of T cells in ablated tumor tissue in comparison to non-cryoablated tissue.

OUTLINE:

At the time of standard of care pleural biopsy, patients undergo cryoablation over 30 minutes, then a sample of tissue from the ablated region and a non-ablated (tumor negative control) region are collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults that have been identified at tumor board with high suspicion for mesothelioma and are anticipated to be surgical candidates, as determined/discussed at Mesothelioma Tumor Board

Exclusion Criteria:

* Patients that have a questionable diagnosis of mesothelioma (i.e. there are other potentially more likely considerations in the differential diagnosis) or in patients that would not be expected to be good surgical candidates

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Local tumor infiltration by cytotoxic cluster of differentiation 8 positive (CD8+) cells | After cryoablation of mesothelioma up to 1 year
  Will be tested by cryoablating a small region of tumor at the time of pleural biopsy.
Preponderance of T cells in ablated tumor tissue in comparison to non-cryoablated tissue | Up to 1 year
  Subsequent fluorescence activated cell sorting for cluster of differentiation 4 positive (CD4+) and CD8+ markers will be performed to identify sub-populations of lymphocytes. The counts will be compared using a one-way paired t-test (two samples from each patient; ablated and non-ablated). The isolated cells will be frozen for potential subsequent use (if the hypothesis for the study is true then subsequent profiling of the cells will be performed, such whole exome sequencing (ribonucleic acid-sequencing) and metabolomic profiling).

CONTACTS AND LOCATIONS:
Overall Officials: Neema Jamshidi, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States